CLINICAL TRIAL: NCT02285049
Title: Cross-Cultural of the Validity, Reliability and Interpretability of Thai-version of Urticaria Control Test (UCT)
Brief Title: Cross-Cultural of the Validity, Reliability and Interpretability of Thai-version of Urticaria Control Test
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: Urticaria Control Test
Record Dates: First submitted 2014-10-17; First posted 2014-11-06 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Urticaria
Keywords: Chronic urticaria; Urticaria Control Test
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Urticaria Control Test: * Evaluation by UAS28, PatGA-LS, PhyGA-LS
  * Fill the UCT and DLQI questionnaire
  Interventions: Other: Urticaria Control Test

INTERVENTIONS:
Other: Urticaria Control Test — * The patients get the 1st UAS28 form and four-week appointment to follow up.
  * Collect completed UAS28 assessment, Patient's global assessment of disease severity (PatGA-LS) and Physician's global assessment of disease control (PhyGA-LS)
  * Then patients fill the 1st UCT and DLQI questionnaire by themselves.
  * The patients get the 2nd UAS28 form and four-week appointment to follow up.
  * At the 2nd visit, collect completed UAS28 assessment. Assessment the severity of chronic urticaria symptoms by Patient's global assessment of disease severity (PatGA-LS) and Physician's global assessment of disease control (PhyGA-LS). The patients fill the UCT and DLQI and questionnaire by themselves.

SUMMARY:
Chronic urticaria symptoms commonly fluctuate from day by day. Consequently the clinical presentation of a patient in each visit is not representative of the current disease status. Dermatologists are trying to integrate an evaluation process of each treatment visit regarding both clinical condition and life quality concern. The Urticaria Control Test is the key for a better treatment outcome in a routine management. To translate this questionnaire into Thai is essential in our subject of interest for offering local patients a higher well-being standard. The Thai-version test will encourage enhanced as well as impactful therapeutic options for Thai chronic urticaria patients.

DETAILED DESCRIPTION:
1. Independently adaption of the UCT questionnaire into Thai version by using forward-backward translation by two bilingual translators. The original German version is translated into Thai by two Thai native speakers, then the study team reviews the Thai-version UCT questionnaire for items comprehensibility and integrates the first consensus version which re-translated into German by German native speaker afterwards. The comparison between the backward German version UCT questionnaire and the original UCT is carried out to find out any misconception and mistranslation in the intermediary forward version of questionnaire. The second version will be tested on 15 chronic urticaria patients to detect any misunderstanding points. Finally, this Thai-version of UCT questionnaire will be used to investigate the validity, reliability, interpretability and minimal clinical important difference.
2. To investigate the validity, reliability and interpretability of Thai-version of Urticaria Control Test, the severity of urticaria symptoms will be assessed by investigators and patients using UAS28, Patient's global assessment of disease severity (PatGA-LS), Physician's global assessment of disease control (PhyGA-LS), the UCT and DLQI questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or above
* Diagnosed as chronic urticaria based on "The EAACI/GA(2) LEN/EDF/WAO Guideline: the 2013 revision and update" by dermatologists
* Literate in Thai language and can complete the questionnaire by themselves.

Exclusion Criteria:

* Have other active skin diseases
* Have a psychiatric problem
* Cannot understand the questionnaire by themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were diagnosed as chronic urticaria
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Convergent validity of Thai version of Urticaria Control Test | 4 week
  Compare the relationship among Urticaria Activity Score (UAS28), Patient's global assessment of disease severity (PatGA-LS), Physician's global assessment of disease control (PhyGA-LS), Dermatology Life Quality Index (DLQI) and Thai-version UCT.

SECONDARY OUTCOMES:
Reliability of Thai version of Urticaria Control Test | 4 week
  * Investigate the internal consistency of Thai-version of UCT by using Cronbach's alpha coefficient.
  * Investigate the intraclass correlation coefficient of Thai-version of UCTscores in the patients who had no clinical change and obtained stable scores between 1st and 2nd visits.
Interpretability of Thai version of Urticaria Control Test | 4 week
  - Investigate the Thai-version of UCT cut-off scores between mild, moderate and severe levels of urticaria control
Screening accuracy (Responsiveness to Change) of Thai version of Urticaria Control Test | 4 week
  Investigate the correlation between UAS28 changes and Thai-version of UCT changes between the 1st and 2nd visits.

CONTACTS AND LOCATIONS:
Overall Officials: Kanokwalai Kulthanan, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital Mahidol University, Bangkok, Bangkok, Thailand